CLINICAL TRIAL: NCT04613882
Title: Quantification of the Visual Benefits of Soft Toric Contact Lenses Compared to Soft Spherical Contact Lenses Over a Range of Refractive Astigmatism
Brief Title: Quantification of the Visual Benefits of Soft Toric Contact Lenses Compared to Soft Spherical Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C19-683 (EX-MKTG-116)
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2022-05

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Soft Toric Custom Made contact lenses (Experimental): Subjects will be randomized to wear Soft Toric custom made contact lenses for 30 minutes in one eye with other eye patched.
  Interventions: Device: Soft Toric Custom Made Contact lens; Device: Soft Spherical Contact Lenses; Device: Spectacle Correction
- Soft Spherical Contact Lenses (Active Comparator): Subjects will be randomized to wear soft spherical contact lens for 30 minutes in one eye with other eye patched
  Interventions: Device: Soft Toric Custom Made Contact lens; Device: Soft Spherical Contact Lenses; Device: Spectacle Correction
- Spectacle Correction (Active Comparator): Subjects will be randomized to wear spectacle Correction for 30 minutes in one eye with other eye patched.
  Interventions: Device: Soft Toric Custom Made Contact lens; Device: Soft Spherical Contact Lenses; Device: Spectacle Correction

INTERVENTIONS:
Device: Soft Toric Custom Made Contact lens — Subjects will be randomized to wear soft toric custom made lenses for 30 minutes in one eye with other eye patched.
Device: Soft Spherical Contact Lenses — Subjects will be randomized to wear soft spherical contact lenses for 30 minutes in one eye with other eye patched.
Device: Spectacle Correction — Subjects will be randomized to wear spectacle Correction for 30 minutes in one eye with other eye patched.

SUMMARY:
The aim of this work is to undertake a range of vision-related measures with soft toric contact lenses soft spherical contact lenses and spectacle lens correction across a range of levels of astigmatism.

DETAILED DESCRIPTION:
This will be a randomised, crossover, partially subject-masked (for contact lenses only), non-dispensing study, controlled by cross-comparison.

ELIGIBILITY:
Inclusion Criteria:

-

Subjects will only be eligible for the study if:

1. They are of legal age between 18 and 40 years.
2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They are current wearers of any soft contact lens (i.e. have worn lenses in the last six months).
5. They have refractive ocular astigmatism between 0.00DC and -1.50DC in one or both eyes.
6. They have a spherical component to their ocular refractive error between 0.00 and - 6.00 DS.
7. They could attain at least 0.10 logMAR distance high contrast visual acuity in one eye with the study lenses within the available power range.
8. They can be fitted satisfactorily with both lens types.
9. They own an acceptable pair of spectacles.
10. They agree not to participate in other clinical research for the duration of this study.

Exclusion Criteria:

-

Subjects will not be eligible to take part in the study if:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They have had corneal refractive surgery.
5. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
6. They are pregnant or breastfeeding.
7. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
8. They have an amblyopic eye, in which case only dominant eye will be assessed for that subject.
9. They have an infectious disease (e.g. hepatitis), any immunosuppressive disease (e.g. HIV) or diabetes.
10. They have a history of severe allergic reaction or anaphylaxis.
11. They have taken part in any other contact lens clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Read, Principal Investigator — Eurolens Research
Locations (1):
- Eurolens Research, Manchester, United Kingdom

REFERENCES:
- [Derived] Read M, Morgan P, Maldonado-Codina C, Orsborn G, Vega J, Navascues-Cornago M. Evaluating the visual benefits of toric soft contact lenses using a novel pupil-controlled vision testing system. Cont Lens Anterior Eye. 2026 Jan 23;49(2):102604. doi: 10.1016/j.clae.2025.102604. Online ahead of print. PMID 41579512

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 59 participants were screened for eligibility. Two participants did not meet the inclusion criteria and therefore were not included in the randomization. Each of the 3 interventions were subdivided into 7 cylinder groups based on required astigmatism range. Of the remaining 57 participants, 4 participants were assigned to cylinder groups which were already full and thus they did not receive any of the interventions. The remaining 53 participants completed the study using the three interventions.
Units Other Than Participants: Eyes
Groups:
- Spherical Contact Lens, Spectacle, Toric Contact Lens: Spherical CL for 30 minutes, then Spectacles for 30 minutes, then Toric CL for 30 minutes
- Spherical Contact Lens, Toric Contact Lens, Spectacle: Spherical CL for 30 minutes, then Toric CL for 30 minutes, then Spectacles for 30 minutes
- Spectacle, Spherical Contact Lens, Toric Contact Lens: Spectacles for 30 minutes, then Spherical CL for 30 minutes, then Toric CL for 30 minutes
- Spectacles, Toric Contact Lens, Spherical Contact Lens: Spectacles for 30 minutes, then Toric CL for 30 minutes, then Spherical CL for 30 minutes
- Toric Contact Lens, Spherical Contact Lens, Spectacles: Toric CL for 30 minutes, then Spherical CL for 30 minutes, then Spectacles for 30 minutes
- Toric Contact Lens, Spectacles, Spherical Contact Lens: Toric CL for 30 minutes, then Spectacles for 30 minutes, then Spherical CL for 30 minutes
Period: First Intervention
Arm/Group | Spherical Contact Lens, Spectacle, Toric Contact Lens | Spherical Contact Lens, Toric Contact Lens, Spectacle | Spectacle, Spherical Contact Lens, Toric Contact Lens | Spectacles, Toric Contact Lens, Spherical Contact Lens | Toric Contact Lens, Spherical Contact Lens, Spectacles | Toric Contact Lens, Spectacles, Spherical Contact Lens
Started | 14; 23 Eyes | 6; 9 Eyes | 9; 15 Eyes | 5; 6 Eyes | 6; 9 Eyes | 13; 22 Eyes
Completed | 14; 23 Eyes | 6; 9 Eyes | 9; 15 Eyes | 5; 6 Eyes | 6; 9 Eyes | 13; 22 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes
Period: Second Intervention
Arm/Group | Spherical Contact Lens, Spectacle, Toric Contact Lens | Spherical Contact Lens, Toric Contact Lens, Spectacle | Spectacle, Spherical Contact Lens, Toric Contact Lens | Spectacles, Toric Contact Lens, Spherical Contact Lens | Toric Contact Lens, Spherical Contact Lens, Spectacles | Toric Contact Lens, Spectacles, Spherical Contact Lens
Started | 14; 23 Eyes | 6; 9 Eyes | 9; 15 Eyes | 5; 6 Eyes | 6; 9 Eyes | 13; 22 Eyes
Completed | 14; 23 Eyes | 6; 9 Eyes | 9; 15 Eyes | 5; 6 Eyes | 6; 9 Eyes | 13; 22 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes
Period: Third Intervention
Arm/Group | Spherical Contact Lens, Spectacle, Toric Contact Lens | Spherical Contact Lens, Toric Contact Lens, Spectacle | Spectacle, Spherical Contact Lens, Toric Contact Lens | Spectacles, Toric Contact Lens, Spherical Contact Lens | Toric Contact Lens, Spherical Contact Lens, Spectacles | Toric Contact Lens, Spectacles, Spherical Contact Lens
Started | 14; 23 Eyes | 6; 9 Eyes | 9; 15 Eyes | 5; 6 Eyes | 6; 9 Eyes | 13; 22 Eyes
Completed | 14; 23 Eyes | 6; 9 Eyes | 9; 15 Eyes | 5; 6 Eyes | 6; 9 Eyes | 13; 22 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Population: There are six reporting groups for each of the randomization sequences of three study interventions. Here, we are not considering participants as some of the participants had only one eye examined and some of the participants had two eye examined. Therefore, we take number of eyes into consideration for better understanding and accuracy.
Units Other Than Participants: Eyes
Groups:
- Spherical Contact Lens, Spectacles, Toric Contact Lens: Spherical CL for 30 minutes, then Spectacles for 30 minutes, then Toric CL for 30 minutes
- Spherical Contact Lens, Toric Contact Lens, Spectacles: Spherical CL for 30 minutes, then Toric CL for 30 minutes, then Spectacles for 30 minutes
- Spectacles, Spherical Contact Lens, Toric Contact Lens: Spectacles for 30 minutes, then Spherical CL for 30 minutes, then Toric CL for 30 minutes
- Total: Total of all reporting groups
Arm/Group | Spherical Contact Lens, Spectacles, Toric Contact Lens | Spherical Contact Lens, Toric Contact Lens, Spectacles | Spectacles, Spherical Contact Lens, Toric Contact Lens | Spectacles, Toric Contact Lens, Spherical Contact Lens | Toric Contact Lens, Spherical Contact Lens, Spectacles | Toric Contact Lens, Spectacles, Spherical Contact Lens | Total
Number analyzed (Participants) | 14 | 6 | 9 | 5 | 6 | 13 | 53
Number analyzed (Eyes) | 23 | 9 | 15 | 6 | 9 | 22 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (4.8) | 27.3 (5.6) | 25.9 (5.0) | 28.2 (7.7) | 25.4 (6.7) | 27.8 (6.3) | 26.5 (5.7)
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 14 | 5 | 13 | 6 | 3 | 17 | 58
  Male | 9 | 4 | 2 | 0 | 6 | 5 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
    (all) |  |  |  |  |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual acuity was assessed using logMAR for each intervention.
Time Frame: Baseline with low contrast VA
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- Overall Participants: Total participants who completed the study
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
logMAR | 0.2 (0.09)

2. Primary Outcome: Visual Acuity
Description: Visual acuity was assessed using logMAR for each intervention.
Time Frame: After 30 minutes of dispense (Low Contrast VA)
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- Soft Spherical Contact Lenses; Soft Toric Custom Made Contact Lenses; Spectacle Correction: Participants wore a spherical contact lens, a custom-made toric contact lens, and a spectacle correction, each in a random sequence for 30 minutes. Each optical correction was worn in one eye only, with the other eye patched. Participants had either a single eye or both eyes evaluated.
Arm/Group | Soft Spherical Contact Lenses | Soft Toric Custom Made Contact Lenses | Spectacle Correction
Number analyzed (Participants) | 53 | 53 | 53
Number analyzed (Eyes) | 84 | 84 | 84
logMAR | 0.28 (0.013) | 0.24 (0.09) | 0.21 (0.09)

3. Primary Outcome: Visual Acuity
Description: Visual acuity was assessed using logMAR for each intervention.
Time Frame: Baseline with High contrast VA
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
logMAR | -0.07 (0.07)

4. Primary Outcome: Visual Acuity
Description: Visual acuity was assessed using logMAR for each intervention.
Time Frame: After 30 minutes of dispense (High Contrast VA)
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Soft Spherical Contact Lenses | Soft Toric Custom Made Contact Lenses | Spectacle Correction
Number analyzed (Participants) | 53 | 53 | 53
Number analyzed (Eyes) | 84 | 84 | 84
logMAR | -0.02 (0.11) | -0.08 (0.07) | -0.1 (0.06)

5. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Conjunctival Redness
Description: Slit lamp Biomicroscopy findings were assessed on Efron Grading scales scored to the nearest 0.1 on a scale of 0 - 4 (0=normal, 1=trace, 2=mild, 3=moderate, 4=severe).
  The assessments done were recorded prior to the first intervention.
  Here the time frame used is "Entrance" which refers to the time prior to wear of study lens.
Time Frame: Entrance (Prior to wear of study lens)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 1.0 (0.3)

6. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Conjunctival Redness
Description: Slit lamp Biomicroscopy findings were assessed on Efron Grading scales scored to the nearest 0.1 on a scale of 0 - 4 (0=normal, 1=trace, 2=mild, 3=moderate, 4=severe).
  The assessments were done following the removal of the third intervention. Here the time frame used is "Exit" which refers to those measurements taken post-lens/spectacle wear.
Time Frame: At Exit (After 30 minutes in each of three interventions)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 1.0 (0.3)

7. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Limbal Redness
Description: as for outcome 5
Time Frame: Entrance (Prior to wear of study lens)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 0.9 (0.3)

8. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Limbal Redness
Description: as for outcome 6
Time Frame: At Exit (After 30 minutes in each of three interventions)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 0.9 (0.3)

9. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Corneal Staining
Description: as for outcome 5
Time Frame: Entrance (Prior to wear of study lens)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 0.2 (0.5)

10. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Corneal Staining
Description: as for outcome 6
Time Frame: At Exit (After 30 minutes in each of three interventions)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 0.3 (0.5)

11. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Conjunctival Staining
Description: as for outcome 5
Time Frame: Entrance (Prior to wear of study lens)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 0.4 (0.4)

12. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Conjunctival Staining
Description: as for outcome 6
Time Frame: At Exit (After 30 minutes in each of three interventions)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 0.6 (0.5)

13. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Papillary Conjunctivitis
Description: as for outcome 5
Time Frame: Entrance (Prior to wear of study lens)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 1.1 (0.3)

14. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Papillary Conjunctivitis
Description: as for outcome 6
Time Frame: At Exit (After 30 minutes in each of three interventions)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 1.1 (0.3)

15. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Corneal Oedema
Description: as for outcome 5
Time Frame: Entrance (Prior to wear of study lens)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 0.0 (0.0)

16. Secondary Outcome: Slit Lamp Biomicroscopy Findings - Corneal Oedema
Description: as for outcome 6
Time Frame: At Exit (After 30 minutes in each of three interventions)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Participants
Number analyzed (Participants) | 53
Number analyzed (Eyes) | 84
units on a scale | 0.0 (0.0)

ADVERSE EVENTS:
Time Frame: The data was collected in the time frame of 90 days
Description: [Not Specified]
Groups:
- Overall Study: It is not possible to report the adverse Events per intervention as the measurements were taken prior to the first intervention and the following third intervention. Thus, the Adverse Events reporting have been combined. The eye twitch and migraine occurred after wearing all three interventions (Spectacles, Spherical Contact Lens and Toric Contact Lens) and thus these data cannot be subdivided. For the corneal scar and asymptomatic CIE these were observed on study but following wear of their habitual contact lenses and occurred prior to wear of the study interventions and thus these data cannot be further subdivided.
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 4/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=57)
Corneal Scar (Eye disorders) | 1
asymptomatic corneal infiltrate event (Eye disorders) | 1
Twitching in the eye (Eye disorders) | 1
Migraine (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT04613882/Prot_SAP_000.pdf